CLINICAL TRIAL: NCT00116012
Title: A Randomized, Double-Blind Placebo-Controlled Study to Assess the Safety of Factor VIIa/Tissue Factor Inhibitor, Recombinant Nematode Anticoagulant Protein c2 (rNAPc2), in Subjects With Non-ST-Elevation Acute Coronary Syndromes - ANTHEM (Anticoagulation With rNAPc2 to Help Eliminate MACE)/TIMI 32. Amendment #3 - A Single Arm, Open-Label Study of rNAPc2 With Reduced Doses of Unfractionated Heparin
Brief Title: Anticoagulation With rNAPc2 to Eliminate MACE/TIMI 32
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCA Biopharma, Inc. (Industry)
Collaborators: The TIMI Study Group (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NUVO-0201; ANTHEM
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2006-11-29 (Estimated); Status verified 2006-11

CONDITIONS: Coronary Disease
Keywords: acute coronary syndrome; rNAPc2; unstable angina; Non-STE myocardial infarction; ST elevation; cardiac enzymes; acute coronary syndromes; factor VIIa; tissue factor; nematode anticoagulant protein c2; anticoagulants; thrombin inhibitors; thrombosis
MeSH Terms: conditions — Coronary Disease; Acute Coronary Syndrome; Angina, Unstable; Thrombosis | interventions — anti-coagulant protein C2, Ancylostoma caninum

INTERVENTIONS:
Drug: rNAPc2

SUMMARY:
The primary focus of this study is to explore the safety of a range of doses of rNAPc2 in subjects who are managed in hospitals that most typically practice an early invasive strategy (catheterization during the index admission). After completion of the ascending dose-ranging part of the trial and review of these data by the Data and Safety Monitoring Board (DSMB), the maximum tolerated dose of rNAPc2 will be studied in single-arm, open-label panels (approximately 25 subjects each) of rNAPc2 with descending doses of unfractionated heparin (UFH).

DETAILED DESCRIPTION:
Acute coronary syndromes (ACS), which include unstable angina and non-ST-elevation (non-STE) myocardial infarction, represent a serious clinical condition affecting over 1,000,000 people in the US alone. The combined rate of death and myocardial infarction (MI) in ACS patients is 8-15% after one month, in spite of the best current therapy including use of low-molecular weight heparins, glycoprotein IIb/IIIa (GPIIb/IIIa) inhibitors, and an early invasive strategy. Given the high prevalence of the disorder, further improvements in the outcomes in these patients are very desirable.

It is currently believed that the principle cause of the clinical symptoms characterizing ACS results from the transient thrombotic occlusion of one or more coronary vessels. Coronary thrombosis is initiated by the exposure of the protein tissue factor (TF), which can be found in the sub-endothelial layer of the blood vessel and is a major component of atherosclerotic gruel. The exposure of TF following vascular damage or rupture of a coronary atherosclerotic plaque, results in the rapid formation of the enzymatic complex composed of TF and the serine protease factor VIIa (fVIIa/TF). The fVIIa/TF complex initiates an amplified cascade of proteolytic activation steps resulting in the formation of the serine protease thrombin. The highly amplified generation of thrombin localized to the site of vascular damage or plaque rupture, coupled with the high-shear rheological environment of the coronary vessel, results in the activation and subsequent aggregation of platelets and the formation of an insoluble matrix of fibrin resulting in a platelet-rich thrombus.

The critical role of the fVIIa/TF complex in the initiation of coronary thrombosis suggests that it may be an ideal target for inhibitors that will result in an attenuation of thrombin generation and subsequent thrombus formation. Recombinant nematode anticoagulant protein c2 (rNAPc2) is a novel and potent inhibitor of fVIIa/TF that may improve current therapeutic strategies in reducing the extent of coronary thrombosis and subsequent clinical events in patients diagnosed with ACS.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 75 years inclusive
* Ischemic symptoms lasting >= 5 minutes at rest within the prior 48 hours
* Able to be randomized within 48 hours of recent ischemic events
* At least one of the following criteria (A, B, or C): A. Elevation of CK-MB or troponin above upper limit of normal OR B. ST segment deviation (depression or transient elevation) of at least 0.5 mm OR C. TIMI risk score >= 3, defined as three or more of the following:

  * Age >= 65;
  * At least 3 of the following risk factors: hypertension, diabetes mellitus, current smoker (within 1 year), dyslipidemia, family history of premature coronary artery disease (< age 60);
  * Known or prior coronary artery stenosis > 50%;
  * Daily aspirin use for at least 7 days;
  * >= 2 ischemic episodes at rest lasting >= 15 minutes each within the prior 24 hours;
  * Elevation of CK-MB OR troponin above upper limit of normal;
  * ST segment deviation (depression or transient elevation) of at least 0.5 mm.
* Ability to understand and willingness to give written informed consent
* Planned early invasive strategy in the index hospitalization

Exclusion Criteria:

* Index event is ST-segment elevation MI or new LBBB
* CABG is planned within 7 days
* ACS is secondary to non-atherosclerotic mechanism (e.g. thyrotoxicosis, anemia)
* Prior participation in ANTHEM-TIMI 32, prior exposure to rNAPc2, or participation in a study with any experimental drug or device within 30 days
* Pregnancy, lactation or use of an intrauterine device (note: women of childbearing potential must have a negative b-HCG)
* Active renal disease, Cr > 4 mg/dl, or history of renal transplantation
* History of a bleeding diathesis or recurrent bleeding episodes
* Medical comorbidities which place subject at risk for hemorrhage, including, but not limited to, prior cerebral hemorrhage, arteriovenous malformation, non-hemorrhagic CVA or TIA, GI bleed, active PUD, advanced liver or renal disease. Major trauma, surgery, CNS, spinal or eye surgery within 6 months, or parenchymal organ biopsy within 14 days.
* Uncontrolled hypertension (SBP > 180, DBP > 100) despite 1 hour of adequate treatment
* Gross hematuria within 1 month unless catheterized and subsequently resolved
* Chronic warfarin (INR > 1.4) or anticipated therapy for warfarin
* Platelet count < 120,000/mm3 at randomization or history of thrombocytopenia (confirm in a blue-top tube using sodium citrate)
* Significant anemia (M: Hg < 11 g/dL, F: Hg < 10 g/dL) at randomization
* Active liver disease or ALT and AST > 3 x ULN not felt to be part of presenting ACS
* Fibrinolytic agent within 24 hours or planned use of fibrinolytics
* Known allergy or intolerance to aspirin
* Known allergy to heparin, enoxaparin or pork-based products
* History of heparin-induced thrombocytopenia (type 1 or 2)
* Any condition for which the investigator feels enrollment in the study would place the subject at unacceptable risk (e.g. substance abuse)
* Part 2 ONLY: Use of LMWH or Xa inhibitor (e.g. Angiomax, Argatroban) >= 12 hours before randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-06

PRIMARY OUTCOMES:
Evaluation of the effects of a range of doses of rNAPc2 in subjects with non-STE acute coronary syndrome on safety and laboratory parameters from randomization until 7 days after the last dose of study drug

SECONDARY OUTCOMES:
Evaluation of the effects of a range of doses of rNAPc2 on the presence of ischemia following randomization as identified via continuous ST segment (Holter) monitoring
Evaluation of the effects of a range of doses of rNAPc2 on pharmacodynamic and pharmacokinetic measures
Evaluation of the effects of rNAPc2 on major cardiovascular clinical events over the period from randomization until six months following randomization
Assessment of the ability of rNAPc2 to blunt the release of markers of necrosis
Exploration of the relationship between genetic variation and rNAPc2 efficacy
Evaluation of the efficacy and safety of rNAPc2 with reduced-dose (including no) unfractionated heparin (UFH)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deitcher, MD, Study Director — ARCA Biopharma, Inc.
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Giugliano RP, Wiviott SD, Stone PH, Simon DI, Schweiger MJ, Bouchard A, Leesar MA, Goulder MA, Deitcher SR, McCabe CH, Braunwald E; ANTHEM-TIMI-32 Investigators. Recombinant nematode anticoagulant protein c2 in patients with non-ST-segment elevation acute coronary syndrome: the ANTHEM-TIMI-32 trial. J Am Coll Cardiol. 2007 Jun 26;49(25):2398-407. doi: 10.1016/j.jacc.2007.02.065. Epub 2007 Jun 11. PMID 17599602
- See also: Company website — http://www.nuvelo.com